CLINICAL TRIAL: NCT07197047
Title: Neck Static Stretching Acutely Reduces Blood Pressure Through Reduction of Tissue Stiffness: A Randomized Crossover Trial
Brief Title: Neck Static Stretching Acutely Reduces Blood Pressure Through Reduction of Tissue Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Ewan Thomas, Ewan Thomas, Associate Professor in Psychology, Educational Science and Human Movement, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ST-BP 306/2025
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Healthy Participants; Healthy Subjects; Healthy Volunteers; Stretching; Stretch; Static Stretching
Keywords: stretching; static stretching; neck stretching; neck static stretching; blood pressure; systolic blood pressure; diastolic blood pressure; tissue stiffness; heart rate variability; blood

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SS (Experimental): Neck static stretching
  Interventions: Other: Neck static stretching
- CC (No Intervention): Control Condition --> participants sat silently on a chair without performing any stretching intervention

INTERVENTIONS:
Other: Neck static stretching — The static stretching intervention targeted the right posterolateral region of the neck. The stretching protocol consisted of four sets of 45 seconds each, separated by 45-second rest intervals, for a total intervention time of 3 minutes. Seated in a chair, participants performed the stretch by gently flexing their head forward and to the left in an anterolateral direction, using their contralateral (left) hand to assist the movement and ensure selective stretching of the right posterolateral region of the neck. Participants were asked to achieve a subjective discomfort intensity of at least 8 out of 10 on the Numerical Rating Scale (NRS), where 0 represents "no pain" and 10 indicates "the strongest pain imaginable"
  Arms: SS

SUMMARY:
Stretching is usually done to improve flexibility and joint movement. Recent research suggests that stretching may also affect the body's heart and blood vessels. For example, stretching may help lower blood pressure, reduce stress in the nervous system, and improve how flexible or stiff blood vessels are.

Blood pressure is the force of blood pushing against the walls of the arteries. It can change based on how much blood the heart pumps and how tight or relaxed the small blood vessels are. Stretching may help relax these vessels and support the parasympathetic nervous system. This system helps the body stay calm and controls functions like heart rate and blood pressure. From blood pressure values, mean arterial pressure (MAP) can be derived using a standard formula. MAP represents the average arterial pressure across the entire cardiac cycle, encompassing both systole and diastole, and is determined by cardiac output in relation to peripheral vascular resistance, the resistance within the circulatory system that sustains blood pressure, regulates blood flow, and reflects an essential component of cardiac function.

The goal of this study was to test whether a short session of static stretching of the neck can lower blood pressure and MAP in healthy subjects. The investigators also measured tissue stiffness (how firm the tissue is) and heart rate variability (a marker of how the nervous system controls the heart). These measures may help explain why blood pressure and MAP change after stretching.

This study tested the hypothesis that static neck stretching may reduce blood pressure and MAP either by decreasing tissue stiffness, thereby facilitating blood flow through reduced peripheral resistance, or by shifting autonomic balance toward enhanced parasympathetic activity. Should the findings confirm the initial hypothesis of blood pressure and MAP reductions, stretching could represent a simple, practical, and effective strategy to support blood pressure and hémodynamic monitoring.

DETAILED DESCRIPTION:
Participants were recruited from the student population of the University of Palermo.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female participants
* ≥ 18 years old

Exclusion Criteria:

* orthopedic disorders
* neurological disorders
* metabolic disorders
* cardovascular disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Blood pressure was measured two times in each session (SS and CC): once at the beginning (when the participant arrived, T0) and once right after the stretching (SS) or control condition (CC) (T1).
  Investigators measured blood pressure while participants were sitting. A reliable blood pressure machine was used. Participants sat and rested for 5-10 minutes to let their blood pressure settle. The cuff was placed on the bare upper arm, about 2 centimeters above the inside of the elbow, with the arm supported at heart level. During the measurement, participants were asked to sit still, stay relaxed, and not talk. Data will be shown as means with standard deviations. To compare baseline values between SS and CC, investigators will first use paired t-tests. Invesigators will then check the data distribution and apply a repeated measures analysis of variance (two conditions × two time points) to look at the effects of time and condition. In the presence of a significant time × condition interaction, post hoc analyses with Scheffé correction will be conducted to locate the differences. Effect sizes will be calculated and reported as partial eta squared (η²p).
Mean Arterial Pressure | MAP was obtained two times for each session (SS and CC): once at the beginning (baseline, T0) and once right after the stretching (SS) or the control condition (CC) (T1).
  MAP was extrapolated from blood pressure using the following formula: MAP = DP + 1/3(SP - DP). Data will be shown as means with standard deviations. To compare baseline values between SS and CC, investigators will first use paired t-tests. Invesigators will then check the data distribution and apply a repeated measures analysis of variance (two conditions × two time points) to look at the effects of time and condition. In the presence of a significant time × condition interaction, post hoc analyses with Scheffé correction will be conducted to locate the differences. Effect sizes will be calculated and reported as partial eta squared (η²p).

SECONDARY OUTCOMES:
Tissue stiffness | Tissue stiffness was measured two times in each session (SS and CC): once at the beginning (when the participant arrived, T0) and once right after the stretching (SS) or control condition (CC) (T1).
  Tissue stiffness was measured with a small handheld device (NEUTONE TDM-N1, TRY-ALL Corp., Japan). This device gently pressed into the skin with a fixed pressure to see how deep it could go. The bone at the base of the neck (C7) was used as a reference point. Measurements were taken on both sides of this bone, 2 centimeters to the right and left. Participants lay face down on a medical bed and were asked to stay completely relaxed. Data will be shown as means with standard deviations. To compare baseline values between SS and CC, investigators will first use paired t-tests. Invesigators will then check the data distribution and apply a repeated measures analysis of variance (two conditions × two time points) to look at the effects of time and condition. In the presence of a significant time × condition interaction, post hoc analyses with Scheffé correction will be conducted to locate the differences. Effect sizes will be calculated and reported as partial eta squared (η²p).
Heart rate variability and heart rate | Heart rate variabilty and heart rate were measured two times in each session (SS and CC): once at the beginning (when the participant arrived, T0) and once right after the stretching (SS) or control condition (CC) (T1).
  Heart rate (HR) and heart rate variability (HRV) were measured with a Polar H10 chest strap sensor, a device known to give accurate results. To prepare, participants were asked not to drink coffee or alcohol, avoid hard exercise for 24 hours, and keep their normal sleep routine. The tests were always done at the same time of day in both conditions (SS and CC) to avoid daily rhythm effects. Participants lay on their back and rested for 5 minutes before the test. Then, HR and HRV were recorded for another 5 minutes while they breathed normally. The chest strap was placed just below the chest bone and secured around the chest. Once the signal was ready, data were sent automatically to a mobile app (Elite HRV). HRV shows how much the time between heartbeats changes. Average HR was calculated from the same recordings. All data were later analyzed with special software (Kubios HRV). The same approach proposed for the other outcomes will be used for data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol: More Detailed Study Protocol (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT07197047/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis Plan (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT07197047/Prot_SAP_001.pdf